CLINICAL TRIAL: NCT05880394
Title: Somatostatin Receptor Imaging Study of Estrogen Receptor Positive (ER+) Metastatic Breast Cancer
Brief Title: Study of Dotatate Imaging in Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Gary Ulaner, Director of Molecular Imaging and Therapy, Hoag Family Cancer Institute, Hoag Memorial Hospital Presbyterian
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 163-22-CA
Record Dates: First submitted 2023-02-24; First posted 2023-05-30 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Gallium-68 DOTATATE — Gallium-68 DOTATATE is a diagnostic agent for use with positron emission tomography (PET) for localization of somatostatin receptor expression on tumors.
Drug: Copper-64 DOTATATE — Copper-64 DOTATATE is a diagnostic agent for use with positron emission tomography (PET) for localization of somatostatin receptor expression on tumors.

SUMMARY:
This will be a Phase 2 clinical trial to assess somatostatin receptor (SSTR) expression in Stage IV estrogen receptor positive (ER+) breast cancer using Gallium-68 DOTATATE or Copper-64 DOTATATE PET/CT.

DETAILED DESCRIPTION:
Subjects with metastatic breast cancer are planned to be enrolled to undergo Gallium-68 DOTATATE or Copper-64 DOTATATE PET/CT imaging at one time point. SSTR uptake in metastatic lesions will be evaluated by independent central review (ICR). FDG PET and bone scans will also be performed within +/- 3 weeks of DOTATATE imaging.

The primary objective of this study is to evaluate uptake of Gallium-68 DOTATATE or Copper-64 DOTATATE in metastatic ER+ breast cancer lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years at the time of signing the informed consent.
* Biopsy proven, ER+, HER2 any, clinically progressive, Stage IV breast cancer requiring restaging.
* For women of childbearing potential (WOCBP):

  a. Negative serum pregnancy test within 48 hours of Ga-68-DOTATATE injection. A women is considered to be of childbearing potential if she is post-menarchal, has not reached postmenopausal state (≥ 12 continuous months of amenorrhea [no menstrual bleeding of any kind, including menstrual period, irregular bleeding, spotting, etc.] with no identified cause other than menopause), and has not undergone surgical sterilization (total hysterectomy, or bilateral tubal ligation or bilateral oophorectomy at least 6 weeks before taking study drug).
* Willingness and ability to provide written informed consent prior to any study-specific assessments and procedures commence.

Exclusion Criteria:

* Known hypersensitivity to Gallium-68 DOTATATE or Copper-64 DOTATATE, octreotate, or any of the excipients of Gallium-68 DOTATATE or Copper-64 DOTATATE
* Current high-dose glucocorticoid (≥ 20 mg prednisone daily or equivalent); long acting SSA within the last 28 days; short acting SSA that cannot be interrupted for 24 hours.
* Unable to perform PET/CT scans according to technical specifications and local guidelines.
* Concurrent primary malignancy, except adequately treated carcinoma in situ, non-melanoma carcinoma of the skin or any other curatively treated malignancy that has achieved complete response and is not expected to require treatment for recurrence during participation in the study.
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Unable or unwilling to comply with the requirements of the study protocol.
* Prior participation in any interventional clinical study within 30 days prior to SSTR PET/CT scan.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Uptake of Ga-68-DOTATATE or Copper-64 DOTATATE using Krenning Score and standardized uptake value (SUV) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ulaner, MD, PhD, Principal Investigator — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No